CLINICAL TRIAL: NCT03157505
Title: Efficacy and Safety of Birch Pollen Immunotherapy in Local Allergic Rhinitis
Acronym: LARbirch
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Andrzej Bozek, MD PhD, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 605060184JB
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Allergic Rhinitis; Allergic Reaction
MeSH Terms: conditions — Rhinitis, Allergic; Hypersensitivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Purethal Birch immunotherapy (Active Comparator): Purethat Birch intervention and symptomatic treatment for 24 months
  Interventions: Drug: Purethal Birch immunotherapy
- placebo and symptomatic treatment (Placebo Comparator): placebo intervention and symtomatic treatment during 24 months
  Interventions: Other: Placebo and symptomatic treatment

INTERVENTIONS:
Drug: Purethal Birch immunotherapy — Purethal birch was administered as perennial therapy: 24 months
  Other Names: allergen specific immunotherapy
  Arms: Purethal Birch immunotherapy
Other: Placebo and symptomatic treatment — symptomatic treatment including: antihitamine drug, nasal dropps and placebo injection
  Arms: placebo and symptomatic treatment

SUMMARY:
Local allergic rhinitis (LAR) is relatively new disease. The question of effect of allergen specific immunotherapy on LAR is open. The randomized, double blind placebo controlled trial of birch subcutaneous AIT on LAR were performed in twenty eight patients. The therapy was performed during 24 months in proportion 15 patients with AIT and 13 placebo. The primary endpoint was decreased of symptoms medication score (SMS). Additionally monitoring serum specific IgE, specific IgG4 and nasal specific IgE (nsIgE) to Bet v1 and parameters of safety and quality of life were provided.

DETAILED DESCRIPTION:
Local allergic rhinitis (LAR) is still an under diagnosed and under treated disease. It is characterised by local production of IgE during natural exposure to aeroallergens. These patients have negative skin prick tests and serum-specific IgEs but have positive nasal provocation tests for aeroallergens. More than 50% of patients with chronic non-allergic rhinitis may have a problem with lack of LAR diagnosis. Misdiagnosis can lead to mistakes in the treatment as well as inefficiencies.

Besides on only local IgE-mediated reaction, allergen immunotherapy (AIT) could be a potential way of treatment such patients. However, there are only sufficient data that the AIT is effective in allergic rhinoconjunctivitis and asthma to pollens and house dust mites and some animal.

The aim of this study was to assess the safety and efficacy of AIT for birch pollen allergens in patients with local allergic rhinitis and a confirmed birch pollen allergy.

ELIGIBILITY:
Inclusion Criteria:

* well document symptoms of rhinitis during birch pollen season
* positive nasal provocation test to birch
* negative results of skin prick tests to inhalant allergen including: D. pteronyssius, D. farinae, grass pollen, birch, hazel, alder Alternaria, and cat.
* negative results of serum total and allergen specific IgE against mentioned allergens.

Exclusion Criteria:

* diagnosis of bronchial asthma, non-allergic rhinitis (especially senile or vasomotor rhinitis) and severe non-stable diseases. All subjects were required to abstain from anti-allergy drugs and glucocorticoid nasal drops for at least 6 weeks prior to the start of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-01-05 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
area under the curve (AUC) | 24 months
  area under the curve (AUC) for the combined symptom and medication scores (SMS)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Fisher, Study Director — Outpatient Clinic Allergy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rondon C, Romero JJ, Lopez S, Antunez C, Martin-Casanez E, Torres MJ, Mayorga C, R-Pena R, Blanca M. Local IgE production and positive nasal provocation test in patients with persistent nonallergic rhinitis. J Allergy Clin Immunol. 2007 Apr;119(4):899-905. doi: 10.1016/j.jaci.2007.01.006. Epub 2007 Mar 2. PMID 17337294
- [Derived] Bozek A, Kolodziejczyk K, Jarzab J. Efficacy and safety of birch pollen immunotherapy for local allergic rhinitis. Ann Allergy Asthma Immunol. 2018 Jan;120(1):53-58. doi: 10.1016/j.anai.2017.10.009. PMID 29273130